CLINICAL TRIAL: NCT04274205
Title: Influence of Brief Supportive Psychotherapy on Major Adverse Cardiovascular Events, Neutrophil-lymphocytes Ratio and Psychological Symptoms in Acute Coronary Syndrome Patients in Intensive Cardiac Care Unit
Brief Title: Influence of Brief Supportive Psychotherapy on Major Adverse Cardiovascular Events, Neutrophil-lymphocytes Ratio and Psychological Symptoms in Acute Coronary Syndrome in Intensive Cardiac Care Unit
Acronym: Supportive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Hamzah Shatri, Head of Psychosomatic Division, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KET-177/UN2.F1/ETIK/PPM.00.02/
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndrome; Brief Supportive Psychotherapy; Intensive Cardiac Care Unit
Keywords: Brief supportive psychotherapy, acute coronary syndrome, major adverse cardiovascular events, neutrophil-lymphocytes ratio, psychological symptoms
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups Acute coronary syndrome group who got brief psychotherapy in five session in 5 days.. 30 minutes in 1 session Acute coronary syndrome group who did not get brief supportive psychotherapy as control Double opened RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Influence on brief supportive psychotherapy (Active Comparator): Intervention group
  Interventions: Other: Intervention group
- Influence of brief supportive psychotherapy (Active Comparator): Control group
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — Brief supportive psychotherapy
  Other Names: Control group

SUMMARY:
There was no MACE in both groups, but there was stroke-major adverse vascular event lower in brief supportive psychotherapy group. There was neutrophil-lymphocytes ratio change better in brief supportive psychotherapy group and significantly in acute coronary syndrome patients without chronic heart failure or coronary arterial disease, also there was psychological symptom (depression) change better in brief supportive psychotherapy and significantly in acute coronary syndrome patients with chronic heart failure or coronary arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome
* 》 18 years old
* have got pharmacological treatment in cardiology standard with or without anxiolytic drug and had got or had not yet got PCI
* be able to communicate and ready to have interview, fill the questioners and psychotherapy

Exclusion Criteria:

* stroke
* cardiogenic shock at admission time
* psychosis
* reject to involve in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 5 days
  Fatal arrhytmia, recurrent myocardial infarction, cardiogenic shock, death

SECONDARY OUTCOMES:
Neutrophil-lymphocytes ratio | 5 days
  Pre-post measure
Psychological symptoms (Hospital anxiety depression scale) | 5 days
  Pre-post measure

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No